CLINICAL TRIAL: NCT03523039
Title: Hemoadsorption With CytoSorb® in Post-Cardiac Arrest Syndrome: a Pilot Study (The CATCH Trial: Post Cardiac Arrest Therapy With Cytosorb Hemoadsorption)
Brief Title: Hemoadsorption With CytoSorb® in Post-Cardiac Arrest Syndrome
Acronym: CATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Antoine Schneider, Doctor, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ID 2018-00421
Record Dates: First submitted 2018-04-19; First posted 2018-05-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest; Cytokine Hemoadsorption
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemoadsorption (Experimental): Hemoadsorption is performed using a CytoSorb® cartridge.
  Interventions: Device: CytoSorb® Hemoadsorption
- Control (No Intervention): Post-cardiac arrest management will be conducted as per institutional protocols.

INTERVENTIONS:
Device: CytoSorb® Hemoadsorption — The therapy is initiated within 6 hours from randomization and maintained for a minimum of 12 consecutive hours to a maximum of 24 consecutive hours.
  Arms: Hemoadsorption

SUMMARY:
This prospective single-centre randomized control trial aims at evaluating the safety and efficacy of hemoadsorption with CytoSorb® in 40 patients with Post-Cardiac Arrest Syndrome admitted to the ICU.

DETAILED DESCRIPTION:
Patients presenting Post-Cardiac Arrest Syndrome (PCAS) in the 24 hours following their admission in Intensive Care Unit will be randomly assigned either to a control group (standard of care) either to a "Hemoadsorption" group. In the latter, the patient will be connected in the 6 hours following randomization to an extracorporeal circuit, in which a Cytosorb ® cartridge will be placed. The circuit will be set up in hemoperfusion mode. The therapy will take place for a minimum of 12 hours and a maximum of 24 hours. Anticoagulation will be achieved using a regional heparin-protamin regimen.

Blood samples will be collected at randomization, T1 (6 hours post-randomization), T2 (12 hours after randomization), T3 (24 hours after randomization), T4 (48 hours after randomization) and T5 (48 hours after randomization), to assess change in inflammatory cytokine levels.

ELIGIBILITY:
Adult (≥18 years old) patients admitted to the ICU after CA, at risk of PACS as defined by the presence of at least one of the following characteristics (at any time within 24hrs of CA):

* Need for a vasoconstrictor (norepinephrine dose > 0.2 µg/kg/min to maintain MAP > 60-70 mmHg, , or equivalent vasoconstrictor agent) for at least one hour
* Serum lactate level > 6 mmol/l
* Time to ROSC > 25 minutes

Exclusion Criteria:

* Evidence for patient's refusal to participate in clinical trials
* Non commitment for ongoing medical therapy (imminent withdrawal of care)
* Cardiac arrest caused by hemorrhagic shock
* Contraindications to therapeutic heparinization
* Shock of primary cardiac origin (LVEF <20%)
* Platelet count <20 G/L
* Deep immunosuppression state, as defined by neutrophils <1 G/L or CD4 <200 /mm3
* Pregnancy
* Acute sickle cell crisis
* Refractory cardiac arrest with ECMO implantation
* Need for renal replacement therapy at time of randomization
* Concomitant enrolment in another study
* Non availability of the research team at time of eligibility at time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change in cytokine levels | From baseline (randomization) to 72 hours after randomization
  Plasma levels reduction of the following inflammatory mediators: IL-1β,IL-1Ra, IL-6, IL-8, IL-10 and TNF-α.
Incidence of Treatment-Emergent Adverse Events | From beginning of hemoadsorption to 24 hours after the end of hemoadsorption, incidence of adverse events such as haemorrhagic complications, catheter-insertion related complications and anaphylactoid reactions
  Rate of intervention-related complications

SECONDARY OUTCOMES:
Vasopressor requirements | From baseline (randomization) to 72 hours after randomization
  Including the number of patients with a 50% decrease in the baseline vasopressor dose after 6, 12, 24, 36 and 48 hours, and the % of patients requiring a vasopressor dose increase within 24 hours of baseline
In-hospital mortality | Day 14, 28 and 90 after randomization
  All-cause mortality
Shock reversal | Within 24 hours from randomization
  Percentage of patients with shock reversal shock reversal being defined in the present study as a norepinephrine dose <0.1μg/kg/min to maintain MAP >60-70 mmHg and a serum lactate level ≤2 mmol/L
Sequential Organ Failure Assessment Score (SOFA) | Day 1 to 7 after randomization
  Total Daily SOFA Score. The score ranges from 0 (best outcome) to 24 (worst outcome).
CRP and Procalcitonin Levels | Day 1, 2, 3 after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Schneider, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monard C, Bianchi N, Poli E, Altarelli M, Debonneville A, Oddo M, Liaudet L, Schneider A. Cytokine hemoadsorption with CytoSorb(R) in post-cardiac arrest syndrome, a pilot randomized controlled trial. Crit Care. 2023 Jan 23;27(1):36. doi: 10.1186/s13054-023-04323-x. PMID 36691082